CLINICAL TRIAL: NCT03992924
Title: A Prospective Evaluation of Clinical Impact of Physiology & Optical Coherence Tomography Guided PCI in STEMI Patients Without Undergoing Primary PCI
Brief Title: Physiology & Optical Coherence in STEMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, director of department of cardiology, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FFR-1
Record Dates: First submitted 2019-06-19; First posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Functional Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- angiography-guided PCI (Active Comparator)
  Interventions: Procedure: function or imaging guided PCI
- FFR-guided PCI (Experimental)
  Interventions: Procedure: function or imaging guided PCI
- OCT-guided PCI (Experimental)
  Interventions: Procedure: function or imaging guided PCI

INTERVENTIONS:
Procedure: function or imaging guided PCI — FFR may be good tools to differentiate patients with STEMI who may not need stent implantation from those who need Optical coherence tomography (OCT) can visualize the microstructure of culprit and the OCT characteristics were validated by histology

SUMMARY:
The objective of this study is to prospectively evaluate the outcomes of different treatment pathways using a Physiology & Imaging guided PCI in patients with STMEI.

A multi-centre study that will prospectively enrol consecutive STEMI patients who don't receive primary PCI within 48 hours after symptom onset because of different reasons.

STEMI patients with culprit lesion stenosis between 0%-90% will be included in this study and randomized to angiography-guided, FFR-guided or OCT guided PCI groups.

ELIGIBILITY:
Inclusion Criteria:

- Age ≥18 years STEMI for 7-30 days Have not undergone PCI because: Stabilization in a non-PCI hospital followed by transfer to a tertiary hospital for further evaluation;Previous emergent angio without ballooning or stenting;Previous emergent Thrombus Aspiration without ballooning or stenting;Pharmacoinvasive therapy Stenosis between 0%-90% TIMI flow grad 3

Exclusion Criteria:

- Left main disease or bypass disease Intolerance to a study drug, metal alloys, or contrast media Life expectancy less than one year Previous PCI or CABG history Cardiogenic shock or LVEF<35% Severe renal or hepatic dysfunction, hemodynamic instability >90% stenosis in culprit lesion TIMI flow ≤ grade 2 Planned surgery within 6 months after index procedure Clinical indications of inability to tolerate DAPT for 12 months Inability to provide written informed consent Participation in another trial before reaching the primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
One-year target lesion failure (TLF) | 12 month
  a composite of cardiac death, target vessel myocardial infarction (TV-MI), or clinically indicated target lesion revascularization (TLR).

SECONDARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Events (MACE) | 12 month
  Death from cardiac causes, ARC defined Stent Thrombosis, Non-fatal MI, Clinically driven target vessel revascularization (TVR) or re-hospitalization due to unstable or progressive angina

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, China